CLINICAL TRIAL: NCT02462096
Title: A Feasibility Study of the InterVene ReLeaf Catheter System in the Creation of Tissue Leaflets in the Femoral and/or Popliteal Vein
Brief Title: A Feasibility Study of the ReLeaf Catheter System
Acronym: ReLeaf
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device modification and simplification of procedural steps
Sponsor: Intervene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-0001
Record Dates: First submitted 2015-05-26; First posted 2015-06-03 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2018-03

CONDITIONS: Chronic Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Subject to undergo the ReLeaf study procedure.
  Interventions: Device: ReLeaf

INTERVENTIONS:
Device: ReLeaf — The ReLeaf catheter is expected to enable a physician to create tissue leaflets that, in turn, generate a valve effect in the deep veins of the legs.
  Other Names: Tissue Leaflet Creation, Creation of Valve-like Effect

SUMMARY:
This study is designed to evaluate the safety and technical feasibility of the ReLeaf Catheter System in the creation of one or more tissue leaflets in the femoral and/or popliteal vein in subjects with chronic venous insufficiency and who meet the protocol entry criteria.

DETAILED DESCRIPTION:
The ReLeaf catheter system is intended for the creation of tissue leaflets in the deep veins where existing valve structures are no longer healthy and effectively moving blood.

This study aims to treat subjects with a documented history of symptomatic chronic venous insufficiency in whom compression therapy for at least 6 months, combined with superficial venous and/or perforator surgery have failed to obtain clinical improvement.

This clinical trial is designed to evaluate the safety and technical feasibility of the ReLeaf Catheter System in the creation of one or more tissue leaflets in the femoral and/or popliteal vein in subjects with chronic venous insufficiency and who meet the protocol entry criteria.

ELIGIBILITY:
Inclusion Criteria:

* History of symptomatic chronic venous insufficiency subjects, clinical category CEAP 3 or greater.
* History of failed compression therapy (of at least 6 months), combined with superficial venous or perforator surgery.
* Femoral and/or popliteal venous reflux of ≥ 1.0 seconds.
* Deep system reflux with Kistner classification grade 2 or higher.
* 18 years of age or older at the time of consent.
* Willing and able to sign the Ethics Committee (EC) approved informed consent form.
* Willing to comply with follow-up evaluations and protocols.

Exclusion Criteria:

* In the Investigator's opinion, venous outflow obstruction that would inhibit adequate flow away from valve site.
* Obstructive features in the femoral or popliteal vein below the proposed tissue leaflet creation site, which, in the Investigator's opinion, will not allow for sufficient blood flow to the tissue leaflet creation site.
* Deep venous system intervention within 6 months of consent.
* Obstructive features or irregularly small luminal diameter in the femoral vein which, in the opinion of the Investigator, will prohibit access to a tissue leaflet creation site.
* Prior deep vein valve surgical intervention in the ipsilateral limb.
* Ankle arthrodesis with secondary muscle atrophy or severely limited ambulation.
* Limb-threatening circulatory compromise.
* Contraindications to anticoagulation therapy that cannot be medically controlled.
* History of symptomatic pulmonary embolism.
* Acute venous thromboembolism within 3 months of consent.
* Comorbidity risks which, in the opinion of the Investigator, limit longevity or likelihood of complying with protocol follow up.
* General contraindications to surgery or the use of anesthesia.
* Uncontrolled heart failure, or NYHA Class III or IV heart failure.
* Open Cardiac surgery (e.g. ventriculotomy, atriotomy) within the past 6 months of consent (Interventional procedures such as stenting or PTCA do not apply.)
* Chronic Kidney Disease with creatinine level of 2mg/dL or higher.
* Active systemic infection or sepsis.
* Pregnant or lactating (positive pregnancy test, women of childbearing potential must be tested).
* Appropriate vascular access is precluded.
* Subject is enrolled in any other clinical study that, in the opinion of the Investigator, may conflict with this study or compromise study results.
* Subject is considered at high risk for non-compliance with the protocol (e.g., inaccessible for follow-up).
* Other invasive surgical procedure within the last 90 days that in the Investigator's opinion would interfere with the study procedure or results.
* History of stroke within the last 6 months.
* Subject is incarcerated or will be incarcerated during the course of the study.
* Untreated significant superficial venous incompetence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2016-10-08 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Technical Feasibility | Day 0
  Technical feasibility will be evaluated as the ability of the ReLeaf Catheter System to access the target site and successfully modify tissue as confirmed by, and in the opinion of, the Investigator. Successful target site access and confirmed tissue modification will be used as a measure of technical feasibility.
Safety (The number of SAEs directly attributable to the study device will be used as a measure of safety) | Day 30
  Safety will be evaluated as freedom from serious adverse events directly attributed to the investigational device. The number of SAEs directly attributable to the study device will be used as a measure of safety.

OTHER OUTCOMES:
Subsequent Efficacy of Treatment | Day 365
  Subsequent efficacy of the treatment following successful creation of the tissue leaflet(s). This will be measured through an assessment of tissue leaflet creation and the tissue leaflets ability to impact blood flow over the course of time.
Durability | Day 365
  Long-term durability of the tissue leaflet(s). Confirmation of tissue leaflet existence over time will be used to assess the durability of the tissue leaflet.
Long-term Safety (Long-term safety will be measured by freedom from SAEs directly attributable to the study device) | Day 365
  Further long-term safety data will be collected, analyzed and reported through the end of the study. Long-term safety will be measured by freedom from SAEs directly attributable to the study device.

CONTACTS AND LOCATIONS:
Locations (1):
- Auckland City Hospital, Auckland, New Zealand